CLINICAL TRIAL: NCT02376387
Title: Evidence Based Evaluation and Acceptance of Donor Hearts for Transplantation
Acronym: DHS
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Oregon Health and Science University (Other); Kaiser Permanente (Other); California Transplant Donor Network (Network); Donor Network of Arizona (Unknown); Gift of Life (Other); Gift of Hope (Other); LifeLink (Industry); New England Organ Bank (Unknown); Life Gift Organ Donation (Unknown); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Kiran Khush, Assistant Professor of Medicine, Stanford University
Other Study IDs: NIH 41169
Record Dates: First submitted 2015-02-17; First posted 2015-03-03 (Estimated); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Heart Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The proposed research will provide evidence-based strategies for the evaluation and acceptance of donor hearts for transplantation. This is relevant to public health because judicious expansion of donor hearts used for transplantation will make this life-saving procedure available to a larger number of patients living with end-stage heart disease.

DETAILED DESCRIPTION:
The demand for donor hearts for transplantation far outstrips the supply; however, only one in three available cardiac grafts are used for transplantation. There are many reasons for graft non-use, but previous studies have failed to demonstrate consistent associations between donor characteristics, donor cardiac function, and adverse recipient outcomes. Thus, there is a critical need to standardize how cardiac allografts are evaluated and accepted for transplantation. The investigators long-term goal is to safely expand the use of available cardiac allografts without adversely affecting transplant recipient outcomes. The investigators propose to carefully characterize the current population of cardiac organ donors, particularly with regards to allograft function; to examine how decisions are made regarding graft acceptance for transplantation; and to systematically evaluate associations between donor characteristics and recipient outcomes. The investigators central hypothesis is that acceptable allografts for heart transplantation are being unnecessarily discarded, and the establishment of an evidence-based process for cardiac donor evaluation and acceptance will increase graft utilization rates while maintaining excellent clinical outcomes. In response to this need, the investigators propose a collaborative study with seven organ procurement organizations representing geographically diverse regions of the United States, to address the following specific aims: (1) To identify clinical correlates of graft function in potential donors being evaluated for heart transplantation. An existing online donor research database will be expanded for standardized collection of data on detailed donor characteristics, especially as pertains to cardiac allograft function. The investigators will perform expert core review of donor echocardiograms, including serial echocardiograms in donors with cardiac allograft dysfunction. Serial electrocardiograms and cardiac biomarkers (Troponin I and B-type natriuretic peptide) will also be studied; (2) To prospectively study reasons for cardiac allograft non-utilization for heart transplantation. Real-time data will be collected on specific reasons for allograft non-acceptance for transplantation in order to study graft acceptance practices and variation in graft utilization nationwide; and (3) To prospectively study associations between donor characteristics and recipient outcomes after heart transplantation. Data will be collected on recipient post-transplant length of hospitalization and survival to identify associations between donor predictors and recipient outcomes. This proposal is innovative because it focuses on an entirely different approach to donor-based research, thereby surmounting the limitations of prior investigations. Completion of the proposed study will have a positive impact by defining how to optimize the evaluation and use of available grafts for heart transplantation, thereby safely expanding the donor pool and increasing the number of heart transplants performed nationwide.

ELIGIBILITY:
Inclusion Criteria:

1. Brain dead (beating heart)
2. 18-65 years of age
3. HIV (-)
4. Donors authorized for research

Exclusion Criteria:

1. Donors not authorized for research
2. HIV (+)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Brain dead donors for heart transplant
Sampling Method: Non-Probability Sample
Enrollment: 4333 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2020-05-26 (Actual); Study Completion 2020-05-26 (Actual)

PRIMARY OUTCOMES:
Donor left ventricular ejection fraction, troponin, BNP, EKG changes (arrhythmias, QT prolongation, repolarization abnormalities, LVH, Q waves) | 5 years
  To identify clinical correlates of cardiac function in potential donors being evaluated for heart transplantation.
Identify decline codes for donor hearts not accepted for transplant | 5 years
  To prospectively study reasons for non-acceptance of hearts offered for transplantation.
Create a statistical tools (e.g. risk prediction model) for donor heart acceptance | 5 years
  To develop clinical tools to assist transplant centers with real-time decisions regarding donor heart acceptance.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Donor Network of Arizona, Phoenix, Arizona
  - California Transplant Donor Network, Oakland, California
  - Kaiser Permanente, San Francisco, California
  - Stanford University, Stanford, California
  - LifeLink, Norcross, Georgia
  - Gift of Hope, Itasca, Illinois
  - New England Organ Bank, Waltham, Massachusetts
  - Gift of Life, Ann Arbor, Michigan
  - Oregon Health and Science University, Portland, Oregon
  - LifeGift, Houston, Texas

REFERENCES:
- [Background] Khush KK, Menza R, Nguyen J, Zaroff JG, Goldstein BA. Donor predictors of allograft use and recipient outcomes after heart transplantation. Circ Heart Fail. 2013 Mar;6(2):300-9. doi: 10.1161/CIRCHEARTFAILURE.112.000165. Epub 2013 Feb 7. PMID 23392789
- [Background] Shah MR, Starling RC, Schwartz Longacre L, Mehra MR; Working Group Participants. Heart transplantation research in the next decade--a goal to achieving evidence-based outcomes: National Heart, Lung, And Blood Institute Working Group. J Am Coll Cardiol. 2012 Apr 3;59(14):1263-9. doi: 10.1016/j.jacc.2011.11.050. PMID 22464255
- [Background] Chen JM, Sinha P, Rajasinghe HA, Suratwala SJ, McCue JD, McCarty MJ, Caliste X, Hauff HM, John R, Edwards NM. Do donor characteristics really matter? Short- and long-term impact of donor characteristics on recipient survival, 1995-1999. J Heart Lung Transplant. 2002 May;21(5):608-10. doi: 10.1016/s1053-2498(01)00367-9. PMID 11983553
- [Background] De La Zerda DJ, Cohen O, Beygui RE, Kobashigawa J, Hekmat D, Laks H. Alcohol use in donors is a protective factor on recipients' outcome after heart transplantation. Transplantation. 2007 May 15;83(9):1214-8. doi: 10.1097/01.tp.0000261713.24244.ea. PMID 17496538
- [Background] Lima B, Rajagopal K, Petersen RP, Shah AS, Soule B, Felker GM, Rogers JG, Lodge AJ, Milano CA. Marginal cardiac allografts do not have increased primary graft dysfunction in alternate list transplantation. Circulation. 2006 Jul 4;114(1 Suppl):I27-32. doi: 10.1161/CIRCULATIONAHA.105.000737. PMID 16820584
- [Background] Nixon JL, Kfoury AG, Brunisholz K, Horne BD, Myrick C, Miller DV, Budge D, Bader F, Everitt M, Saidi A, Stehlik J, Schmidt TC, Alharethi R. Impact of high-dose inotropic donor support on early myocardial necrosis and outcomes in cardiac transplantation. Clin Transplant. 2012 Mar-Apr;26(2):322-7. doi: 10.1111/j.1399-0012.2011.01504.x. Epub 2011 Oct 10. PMID 21981698
- [Background] Patel ND, Weiss ES, Nwakanma LU, Russell SD, Baumgartner WA, Shah AS, Conte JV. Impact of donor-to-recipient weight ratio on survival after heart transplantation: analysis of the United Network for Organ Sharing Database. Circulation. 2008 Sep 30;118(14 Suppl):S83-8. doi: 10.1161/CIRCULATIONAHA.107.756866. PMID 18824775
- [Background] Smits JM, De Pauw M, de Vries E, Rahmel A, Meiser B, Laufer G, Zuckermann A. Donor scoring system for heart transplantation and the impact on patient survival. J Heart Lung Transplant. 2012 Apr;31(4):387-97. doi: 10.1016/j.healun.2011.11.005. Epub 2011 Dec 16. PMID 22177692
- [Background] Weiss ES, Allen JG, Kilic A, Russell SD, Baumgartner WA, Conte JV, Shah AS. Development of a quantitative donor risk index to predict short-term mortality in orthotopic heart transplantation. J Heart Lung Transplant. 2012 Mar;31(3):266-73. doi: 10.1016/j.healun.2011.10.004. Epub 2011 Nov 16. PMID 22093382
- [Background] Wever Pinzon O, Stoddard G, Drakos SG, Gilbert EM, Nativi JN, Budge D, Bader F, Alharethi R, Reid B, Selzman CH, Everitt MD, Kfoury AG, Stehlik J. Impact of donor left ventricular hypertrophy on survival after heart transplant. Am J Transplant. 2011 Dec;11(12):2755-61. doi: 10.1111/j.1600-6143.2011.03744.x. Epub 2011 Sep 11. PMID 21906259